CLINICAL TRIAL: NCT03130504
Title: The Use Of Intramuscular Hydroxyprogesterone Caproate For Management Of Placenta Previa Before 34 Weeks Of Gestation
Brief Title: Intramuscular Hydroxyprogesterone Caproate and Placenta Previa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMHC
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 17α hydroxy progesterone caproate group (Active Comparator)
  Interventions: Drug: 17α hydroxy progesterone caproate
- No intervention group (No Intervention)

INTERVENTIONS:
Drug: 17α hydroxy progesterone caproate — where patients will have a 17α hydroxy progesterone caproate intramuscular injection every week starting from 24 weeks of gestation till completed 37 weeks
  Arms: 17α hydroxy progesterone caproate group

SUMMARY:
Antepartum hemorrhage is defined as bleeding from or within the female genital tract, occurring from 24+0 weeks of pregnancy and till delivery of the fetus. Antepartum hemorrhage occurs in 3-5% of pregnancies and is an important cause of perinatal and maternal morbidity and mortality worldwide.

Placenta previa is a placenta inserted wholly or in part into the lower segment of the uterus. It is classified by ultrasound to Placenta previa major degree when the lower edge of the placenta lies within 2 cm from the internal cervical os and Placenta previa minor degree if the lower edge of the placenta at lower uterine segment but more than 2 cm from internal os. Placenta previa is responsible for 0.03% of maternal mortality and 8.1% of perinatal mortality of 8.1% in the developed world and much more in developing countries.

Many studies in literature proved the positive correlation between the Placenta previa and preterm uterine contractility and also reported that large proportion of women who have Placenta previa associated with vaginal bleeding will have subclinical uterine contractions before the onset of evident vaginal bleeding.

There are many tocolytic agents may have a role in conservative management of Placenta previa such as magnesium sulfate and β-sympathomimetics .Progesterone is essential for continuation of pregnancy and helps in maintenance of pregnancy . Delaying delivery may reduce the fetal morbidity by helping maturity of vital organs. In 2003 Meis et al. in a large randomized placebo-controlled trial found a significant reduction in recurrent preterm birth before 37 weeks for women who received 17αHP-C versus a control group receiving placebo (36.3% versus 54.9%).

ELIGIBILITY:
Inclusion Criteria:

1. Estimated gestational age is ranging between 24 weeks and 26 week's gestation
2. Singleton pregnancy.
3. Placenta previa; either major or minor degrees.
4. Placenta previa with minimal vaginal bleeding or haven't any vaginal bleeding.
5. For outpatient follow ups, women should be living in a nearby area to make follow-up and early transportation are reasonably possible.
6. Accepting to participate in the study.

Exclusion Criteria:

1. Definite rupture of membranes.
2. Established preterm labor.
3. Severe attack of bleeding requiring an immediate intervention.
4. Fetal heart rates instability or non reassuring
5. Intrauterine fetal death or major fetal anomalies.
6. If associated with abruptio placentae
7. Patients with known bleeding disorders or on anticoagulant therapy
8. Patents with severe medical disorders as preeclamptic toxemia, diabetes mellitus, hepato-renal impediment …etc
9. The presence of reported side effects in the mother from 17α hydroxy progesterone caproate like hypersensitivity reactions, cough, dyspnea, and diabetes.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
number of women delivered before 37 weeks | 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No